CLINICAL TRIAL: NCT00209300
Title: Pentasa Once Daily in Ulcerative Colitis for Maintenance of Remission. A European Multi-centre Investigator Blinded Randomized Controlled Study of Pentasa Sachet Comparing One Gram Twice With Two Grams Once Daily
Brief Title: Pentasa Once Daily in Ulcerative Colitis for Maintenance of Remission
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: FE999907 CS003; 2004-004565-15
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis for Maintenance of Remission
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pentasa

SUMMARY:
This is a multi-centre, randomised, controlled, investigator blinded study. The randomisation will be done centrally. The patients will be treated for 1 year, with clinical and laboratory assessments at 0, 4, 8 and 12 months.

Endoscopic examination is at enrollment and on completion of the study (at relapse or after 12 months).

Number of Subjects (Planned and Analysed):

* 360 patients for demonstration of non-inferiority between once daily and twice daily;
* 326 to be analysed in per-protocol (PP) analyses; and
* 360 in intention-to-treat (ITT) analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have an established diagnosis of ulcerative colitis and are in clinical remission with an UC-DAI < 2 at enrollment
2. Extension of the disease > 15 cm distance from anal verge
3. Patients who have had a clinical relapse within the past year. Clinical relapse is defined as activity of the disease for which maintenance therapy had to be adjusted.
4. Patients on oral mesalazine maintenance therapy ≤ 2.5 grams per day
5. 18 years or older
6. Signed informed consent

Exclusion Criteria:

1. Patients with evidence of other forms of inflammatory bowel disease, idiopathic proctitis or infectious disease
2. Patients allergic to acetylsalicylic acid and other salicylate derivates aspirin or salicylates derivatives
3. Patients who used mesalazine > 2.5 grams orally in the previous month,
4. Patients who used rectal mesalazine > 3 grams per week in the previous month
5. Use of corticosteroids (oral and/or rectal routes) within the last month
6. Intake of immunosuppressants within the last 3 months
7. Patients with (known) significant hepatic (up to 2 x upper limit of normal) or (known) renal function abnormalities, to 1.5 x upper limit of normal values
8. Patients with history or physical examination findings indicative of active alcohol or drug abuse
9. Patients with a history of disease, including mental/emotional disorders, that would interfere with their participation in the study
10. Women who are pregnant or nursing (non-menopausal women who are sexually active and do not use effective contraceptives, as judged by the investigator, must have a negative pregnancy test)
11. Patients who participated in another clinical study in the last 3 months
12. Patients who were previously participating in this study
13. Patients with any other disease that may influence the study assessment, such as malignant disease, etc.
14. Patients who are unable to comply with any requirements of the protocol
15. Patients who are unable to write or read local language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2005-05; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (68):
- Belgium (7):
  - UMC Sint-Pieter, Brussels
  - Hôpital Erasme Unité de Recherche, Clinique Gastro-entérologie, Brussels
  - UZ Gent, Ghent
  - UZ Gasthuisberg, Leuven
  - CHR de la Citadelle, Liège
  - Heilig Hart Ziekenhuis, Roeselaere
  - AZ St. Augustinus, Wilrijk
- Czechia (10):
  - Internal department Hospital Tábor, Jaroše
  - Internal department, Hospital Jičín, Jičín
  - Internal department Hospital Chomutov, Kochova
  - Hospital Mladá Boleslav - Internal Department, Mladá Boleslav
  - Gastroenterologie MUDr.V.Abrahámová, Poděbrady
  - Internal department, Hospital of Merciful sisters, Prague
  - Gastroenterological Centre, University Hospital of Charles University, Prague
  - EGK s.r.o, Gastroenterology, Prague
  - Internal department University Hospital Na Bulovce, Prague
  - Internal department Hospital, Příbram
- Denmark (8):
  - Amager Hospital Medicinsk Center, Copenhagen S
  - Helsingor Sygehus, Elsinore
  - Amtsygehuset i Gentofte, Hellerup
  - Sygehus Vendsyssel, Hjørring
  - Naestved Sygehys, Næstved
  - Sonderborg Sygehus, Sønderborg
  - Vejle Sygehus, Vejle
  - Viborg Sygehus, Viborg
- North Karelia Central Hospital, Joensuu, Finland
- Germany (29):
  - Gemeinschaftspraxis Dres. Lupberger, Kraus, Graf Finck von Finckenstein, Augsburg
  - Kreiskrankenhaus Beeskow, Beeskow
  - Gemeinschaftspraxis, Berlin
  - Praxisgemeinschaft für Innere Med./Gastro Dres. med M.-E. v. Gynz-Rekowski & R. Drossel, Berlin
  - Universitätsklinikum Charité, Campus Virchow Klinikum, Berlin
  - St. Josef-Hospital, Bochum
  - Universitätsklinikum Carl-Gustav-Carus, Medizinische Klinik und Poliklinik I, Bonn
  - Gemeinschaftspraxis Dres. Toermer / Boedler, Cologne
  - Gemeinschaftspraxis Dres. Landry, Wilhelm, Bourgeois, Pfeifer, Leibold-Lamprecht, Kindermann, Müller, Dachau
  - Gemeinschaftspraxis, Dinkelsbühl
  - Gemeinschaftspraxis Dres. Weber/Berghaus, Dortmund
  - Universitätsklinikum Carl-Gustav-Carus, Medizinische Klinik und Poliklinik I, Dresden
  - Gemeinschaftspraxis Dres. Zeus/Schenk, Erlangen
  - Medizinische Klinik 1, Frankfurter Diakonie-Kliniken, Markus Krankenhaus, Frankfurt a.M.
  - Facharzt für Innere Medizin / Gastroenterologie, Görlitz
  - Gemeinschaftspraxis, Hamburg
  - Med. Hochschule Hannover, Zentrum Innere Medizin, Hanover
  - Gemeinschaftspraxis Dres. Lupberger, Kraus, Graf Finck von Finckenstein, Hof
  - Gemeinschaftspraxis, Homberg (Efze)
  - Gastroenterologische Gemeinschaftspraxis Dres. Lütke/Weismüller, Koblenz
  - Gemeinschaftspraxis Dres. Dietel/Klugmann, Leipzig
  - Klinikum Leverkusen Medizinische Klinik 2, Leverkusen
  - Gemeinschaftspraxis Dres. Kocjan / Muser, Lüdenscheid
  - Universitätsklinikum Charité, Magdeburg
  - Gemeinschaftspraxis, Mainz
  - Gemeinschaftspraxis Dres. Bokemeyer/Roggel/Kamp, Minden
  - Praxisklinik Dr. Eimiller/Prof. Kellner, München
  - Klinkum rechts der Isar der TUM, München
  - Gemeinschaftspraxis Dres. Kardalinos/Petry, Stuhr / Brinkum
- Netherlands (5):
  - Academisch Medisch Centrum, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - Ziekenhuisgroep Twente, loc. streekziekenhuis Midden-Twente, Hengelo
  - Isala klinieken, JW Zwolle
  - Ikazia ziekenhuis, Rotterdam
- Norway (2):
  - Ullevål Universitetssykehus HF, Oslo
  - Aker universitetssykehus HF, Oslo
- Sweden (6):
  - Centralsjukhuseet Kristianstad Medicinkliniken, Kristianstad
  - Ljungby Lasarett, Ljungby
  - Endoskopienheten Lakarhuset Hoterget, Stockholm
  - Södersjukhuset SöS Medicinkliniken, Stockholm
  - Karolinska Universitetssjukhuset, Stockholm
  - Täby Närsjukhus, Täby